CLINICAL TRIAL: NCT07142304
Title: IMPACT: A Clinical Investigation on IMproving Peripheral Neuropathy Induced by Chemotherapy With Advanced Compression Technology - A Safety and Efficacy Study
Brief Title: The Lilac Device Trial
Acronym: IMPACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luminate Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CLIN-53
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-08

CONDITIONS: Chemotherapy Induced Peripheral Neuropathy (CIPN)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Device: The Lilac Device
- Control (Sham Comparator)
  Interventions: Device: Sham device

INTERVENTIONS:
Device: The Lilac Device — The Lilac Glove and Boot devices are wearable, non-sterile device for patients undergoing cancer treatment who wish to reduce the risk of peripheral neuropathy. Treatment with the Lilac Glove and Boot devices is administered by the healthcare professional in the healthcare environment. The Lilac Glove and Boot devices are designed for continual use; the devices must be fitted and turned on before infusion begins; the devices must be used without interruption during infusion, and for up to two (2) hours after infusion is complete.
  Arms: Treatment
Device: Sham device — The sham device will look, appear to function and worn for the same duration as the Lilac Device. The only difference between the devices is the level of compression applied.
  Arms: Control

SUMMARY:
Chemotherapy drugs, used in the treatment of cancer, have the potential of inducing peripheral neuropathy (PN) as a side effect. This side effect is commonly referred to as CIPN, or chemotherapy-induced peripheral neuropathy.

The Lilac Glove and Boot devices apply a low pressure across the surface of the hands and feet, respectively, to reduce access of chemotherapy to the peripheral nerves on the hands and feet. The small amount of pressure reduces the level of chemotherapy reaching the peripheral nerves, hence increasing the likelihood of nerve preservation during treatment and thus may potentially temporarily prevent the onset of moderate to severe PN symptoms induced by chemotherapy in the hands and feet while receiving treatment

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this clinical investigation, participants must meet ALL the following criteria:

1. Adults ≥ age 18 with diagnosed solid tumor cancer, who have been deemed appropriate for neo-adjuvant or adjuvant chemotherapy.
2. Planned intravenous treatment with at least 4 cycles of chemotherapy, with no planned treatment pause for surgery,

   * With one of the following treatments:

     * Chemotherapy regimens based on Oxaliplatin

       * FOLFOX every 2 weeks
       * FOLFIRINOX every 2 weeks
     * Chemotherapy regimens based on single-agent Paclitaxel

       * Paclitaxel weekly
       * Paclitaxel every 3 weeks
     * Chemotherapy regimens based on Paclitaxel + Carboplatin

       * Paclitaxel weekly with Carboplatin weekly/every 3 weeks
       * Paclitaxel every 3 weeks with Carboplatin every 3 weeks
   * Concurrent administration of the chemotherapies listed in the inclusion criteria with or without targeted agents/immunotherapy at standard doses is allowed (such as trastuzumab, pertuzumab, bevacizumab, pembrolizumab or other immune checkpoint inhibitors).
3. Hands and feet size within the specified study sizing range.
4. Plan to complete taxane- or platinum-based chemotherapy in ≤ 12 months.
5. ECOG performance status 0 - 2.
6. Willing and able to sign informed consent.
7. Willing to comply with and tolerate all study procedures including:

   * Wearing the Lilac Glove and Boot devices for the prescribed duration (devices to be fitted before infusion, and worn during infusion and for up to one (1) hours post infusion),
   * Complete all study related questionnaires.
8. Participants must be able to complete participant specific questionnaires in the languages available to the study

Exclusion Criteria:

Participants are not eligible to participate in the clinical trial if they meet ANY of the following criteria:

1. Baseline peripheral neuropathy of any kind as defined by NCI CTCAE v5.0 grade > 0.
2. Prior exposure to neurotoxic chemotherapy in the previous 1 year, counted as the period since the last neurotoxic chemotherapy treatment (e.g., taxanes, platinum agents, vinca alkaloids, or bortezomib).
3. Positive pregnancy test at baseline for participants with child bearing potential, as per standard of care.
4. Known or suspected allergy or hypersensitivity to any component of the Lilac Glove or Boot device that comes into contact with the study participant. Caution: This product contains natural rubber latex, which may cause allergic reactions.
5. Any open wounds, sores, cysts or injury on the participant's hand or on part of the upper arm where the device will be applied or on the participant's feet or part of the lower leg where the device will be applied, which in the opinion of the investigator will not be healed prior to infusion commencing or who in the opinion of the investigator will be inappropriate for inclusion in this study.
6. Clinically significant peripheral arterial ischemia, as per standard of care, in the opinion of the investigator.
7. Untreated or uncontrolled hypertension, as per standard of care.
8. Poorly controlled diabetes, as per standard of care, in the opinion of the investigator.
9. Weight greater than 140 kg at the time of enrollment.
10. An existing history or suspicion of presence of hand or foot metastasis.
11. Use of other investigational devices or active compression/ cryotherapy interventions for CIPN prevention or management during the study.
12. Participants who are receiving neuropathy directed systemic therapies at the time of enrollment, namely, Pregabalin, Gabapentin, Amitriptyline, Nortriptyline, Venlafaxine, Duloxetine.
13. Participants who, in the opinion of the investigator, will be inappropriate for inclusion into this study or will not comply with the requirements of the study.
14. Participants with cognitive impairment, psychiatric conditions, or mobility limitations that would prevent compliance with study procedures (e.g., inability to wear the device, complete questionnaires, or attend follow-up visits).
15. Current participation in a clinical study or within the last 30 days prior to screening that may cause peripheral neuropathy.
16. Participation in this study at an earlier stage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Occurrence of clinically meaningful overall CIPN symptoms at week 12 of treatment | From first chemotherapy and device treatment to 12 weeks post treatment one
  The occurrence of clinically meaningful overall CIPN symptoms is defined as an absolute increase of 5.06 or more points over baseline in the European Organisation for Research and Treatment of Cancer Quality of Life Chemotherapy Induced Peripheral Neuropathy-20 (EORTC QLQ-CIPN20) score (standardized 0 - 100 scale).
Occurrence of clinically meaningful CIPN symptoms in the hands only at week 12 of treatment | From first chemotherapy and device treatment, to 12 weeks post treatment one
  The occurrence of clinically meaningful CIPN symptoms in the hands only is defined as an absolute increase of 9.60 or more points over baseline in the EORTC QLQ-CIPN20 upper extremity subscale score (standardized 0 - 100 scale)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Palomar Medical Center Poway, Poway, California
  - Hialeah Hospital, Hialeah, Florida
  - Hawaii Cancer Care, Honolulu, Hawaii
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - Health Partners Frauenshuh Cancer Center, Minneapolis, Minnesota
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Mercy Health St. Elizabeth Hospital, Youngstown, Ohio
  - Hospital Sisters Health System - St.Vincent & St.Mary's, Green Bay, Wisconsin

IPD SHARING:
Plan to Share IPD: No